CLINICAL TRIAL: NCT03144635
Title: A Prospective Multicenter Observational Study for Characterization of Renal Function G1b CHC Patients With CKD-3 Treated With Grazoprevir Plus Elbasvir
Brief Title: A Study for G1b CHC Patients With CKD-3 Treated With Grazoprevir Plus Elbasvir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyushu University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Norihiro Furusyo, Associate Professor, Department of General Internal Medicine, Kyushu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KULDS-001
Record Dates: First submitted 2017-04-28; First posted 2017-05-09 (Actual); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis C Viral; Chronic Kidney Disease stage3
Keywords: Direct Acting Antivirals; Grazoprevir; Elbasvir
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Grazoprevir plus Elbasvir (Experimental): Grazoprevir 100 mg plus Elbasvir 50 mg per day for 12 weeks.
  Interventions: Drug: Grazoprevir plus Elbasvir

INTERVENTIONS:
Drug: Grazoprevir plus Elbasvir — An oral dose of 100 mg/day of grazoprevir as well as an oral dose of 50 mg/day of elbasvir for 12 weeks.

SUMMARY:
The regimen using grazoprevir plus elbasvir treatment is promising in Japan, because it may safely be used for the elderly patients with renal dysfunction. Grazoprevir and elbasvir are metabolized in the liver and do not require dose-adjustment for patients with renal dysfunction. However, no data related to efficacy and safety of the grazoprevir plus elbasvir treatment for Japanese elderly patients with renal dysfunction (eGFR<60 mL/min/1.73m2) have been reported. Therefore, physicians are at a loss whether or not to treat the patients with renal dysfunction due to no evidence.

The aim of this study is to investigate the improvement of serum endostatin level of Japanese patients with CKD stage 3 after grazoprevir (NS3/4A protease inhibitor) plus elbasvir (NS5A replication complex inhibitor) treatment by a prospective, multicenter cohort study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 20 years or older.
2. Patients positive for HCV RNA for over 6 months and infected with genotype 1b chronic hepatitis C, including compensated cirrhosis.
3. Patients without co-infection of hepatitis B virus.
4. Patients without co-infection of human immunodeficiency virus
5. Patients with moderate chronic kidney disease (CKD stage 3) (eGFR: 30-59 mL/min/1.73m2). A diagnosis of CKD is only confirmed if repeated eGFR tests for at least 90 days.

Exclusion Criteria:

1. Patients with decompensated cirrhosis (Child Pugh B and C)
2. Patients with albumin <3.0 g/dL and platelets <75,000 /μL
3. Patients with autoimmune hepatitis
4. Constant heavy alcohol drinkers (converted to ethanol ≥60 g/day)
5. Patients who have a history of hypersensitivity to grazoprevir and elbasvir
6. Patients who are pregnant females, or females who may become pregnant, or females who are breastfeeding
7. Patients with heart disease that is hard to control (e.g., very recent cardiac infarction, severe heart failure, unstable arrhythmia)
8. Patients who are under medication with drugs listed as contraindication in a package insert of grazoprevir plus elbasvir treatment
9. Patients judged (by the physician in charge of research) to be inappropriate as subjects for the study for any other reasons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norihiro Furusyo, MD, PhD, Principal Investigator — Kyushu University Hospital
Locations (1):
- Kyushu University Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Furusyo N, Ogawa E, Nakamuta M, Kajiwara E, Nomura H, Dohmen K, Takahashi K, Satoh T, Azuma K, Kawano A, Tanabe Y, Kotoh K, Shimoda S, Hayashi J; Kyushu University Liver Disease Study (KULDS) Group. Telaprevir can be successfully and safely used to treat older patients with genotype 1b chronic hepatitis C. J Hepatol. 2013 Aug;59(2):205-12. doi: 10.1016/j.jhep.2013.03.020. Epub 2013 Mar 28. PMID 23542346
- [Background] Ogawa E, Furusyo N, Yamashita N, Kawano A, Takahashi K, Dohmen K, Nakamuta M, Satoh T, Nomura H, Azuma K, Koyanagi T, Kotoh K, Shimoda S, Kajiwara E, Hayashi J; Kyushu University Liver Disease Study(KULDS) Group. Effectiveness and safety of daclatasvir plus asunaprevir for patients with hepatitis C virus genotype 1b aged 75 years and over with or without cirrhosis. Hepatol Res. 2017 Mar;47(3):E120-E131. doi: 10.1111/hepr.12738. Epub 2016 Jun 10. PMID 27142311
- [Background] Ogawa E, Furusyo N, Kajiwara E, Nomura H, Kawano A, Takahashi K, Dohmen K, Satoh T, Azuma K, Nakamuta M, Koyanagi T, Kotoh K, Shimoda S, Hayashi J. Comparative effectiveness and safety study of triple therapy with simeprevir or telaprevir for non-cirrhotic patients with chronic hepatitis C virus genotype 1b infection. J Gastroenterol Hepatol. 2015 Dec;30(12):1759-67. doi: 10.1111/jgh.13016. PMID 26095167

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Grazoprevir Plus Elbasvir
Started | 80
Completed | 0
Not Completed | 80

BASELINE CHARACTERISTICS:
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 80
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 77 [69 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 80
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 80
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 23.3 [20.7 to 25.2]
Albumin [Median (Inter-Quartile Range); unit: g/dL] | 4.0 [3.6 to 4.2]
Aspartate aminotransferase [Median (Inter-Quartile Range); unit: U/L] | 43 [31 to 65]
Alanine aminotransferase [Median (Inter-Quartile Range); unit: U/L] | 34 [24 to 56]
Gamma-glutamyl transpeptidase [Median (Inter-Quartile Range); unit: U/L] | 35 [19 to 71]
alpha-fetoprotein [Median (Inter-Quartile Range); unit: ng/mL] | 4.3 [3.0 to 12.0]
Cirrhosis [Count of Participants; unit: Participants] | 31
HCV RNA level [Median (Inter-Quartile Range); unit: logIU/mL] | 6.2 [5.9 to 6.6]
Treatment Naive [Count of Participants; unit: Participants] | 69
HCV NS5A RAS [Count of Participants; unit: Participants] — We identified the following as amino-acid resistance-associated substitutions (RAS) to non-structual 5A (NS5A) inhibitor by direct sequencing: NS5A gene amino acid positions 30, 31, and 93 for patients infected with HCV were examined at baseline.
  Participants | 16

OUTCOME MEASURES:

1. Primary Outcome: Change of Serum Endostatin Level (ng/mL) From Baseline to 3 Months
Description: We evaluated the serum endostatin at baseline and 3 months after the treatment initiation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 80
ng/mL
  Baseline | 156 (58)
  3 months | 176 (65)

2. Primary Outcome: Change of eGFR Level (mL/Min/1.73m^2) From Baseline to 3 Months
Description: We evaluated eGFR level at baseline and 3 months after the treatment initiation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 80
mL/min/1.73m^2
  Baseline | 52 (8)
  3 months | 53 (9)

3. Secondary Outcome: Sustained Virological Response-12 (SVR12)
Description: SVR12 was defined as undetectable HCV RNA at week 12 after the end of treatment.
Time Frame: 3 months
Population: Three patients discontinued treatment due to adverse effects.
Measure: Count of Participants; unit: Participants
Groups:
- Intention-to-treat Populations; Per-protocol Populations: Grazoprevir 100 mg plus Elbasvir 50 mg per day for 12 weeks.
  Grazoprevir plus Elbasvir: An oral dose of 100 mg/day of grazoprevir as well as an oral dose of 50 mg/day of elbasvir for 12 weeks.
Arm/Group | Intention-to-treat Populations | Per-protocol Populations
Number analyzed (Participants) | 80 | 77
Participants | 76 | 76

4. Secondary Outcome: Change of Serum Alanine Aminotransferase (ALT) Level (U/L) From Baseline to 3 Months
Description: We evaluated the serum ALT levels at baseline and 3 months after the treatment initiation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 80
U/L
  Baseline | 47 (41)
  3 months | 21 (29)

5. Secondary Outcome: Change of Serum Alpha-fetoprotein Level (ng/mL) From Baseline to 3 Months
Description: We evaluated the serum alpha-fetoprotein levels at baseline and 3 months after the treatment initiation.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 80
ng/mL
  Baseline | 10.7 (17)
  3 months | 4.6 (3.7)

6. Secondary Outcome: Count of Participants With NS3/4A or NS5A Muttations Who Achieved SVR12
Description: We identified the NS3/4A or NS5A muttations by direct sequencing at baseline. Among participants who had mutations, we calcualted the rate of SVR12.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Grazoprevir Plus Elbasvir
Number analyzed (Participants) | 16
Participants | 15

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Grazoprevir Plus Elbasvir
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 3/80
Other Adverse Events (participants affected / at risk) | 0/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Grazoprevir Plus Elbasvir (N=80)
Serious ALT elevation (Hepatobiliary disorders) | 3 — ALT>300 U/L during treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT03144635/Prot_SAP_000.pdf